CLINICAL TRIAL: NCT01442597
Title: Computer Based Training in Cognitive Behavioral Therapy Web-based
Acronym: Man VS Machine
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1004006632; 2P50DA009241-21 (NIH)
Record Dates: First submitted 2011-09-26; First posted 2011-09-28 (Estimated); Last update posted 2020-03-06 (Actual); Status verified 2020-03

CONDITIONS: Substance Abuse
Keywords: cognitive behavior therapy; computer assisted instruction; drug abuse therapy; educational resource design and development
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Individual clinician-provided CBT (Active Comparator): Individual treatment provided by a trained Cognitive Behavioral Therapy (CBT)clinician who will cover the same skills provided by the CBT4CBT computer program.
  Interventions: Behavioral: Individual clinician-provided CBT
- CBT4CBT (Experimental): A computerized program that teaches skills for stopping drug use and increasing coping skills such as how to understand patterns of drug use, coping with cravings, etc.
  Interventions: Behavioral: CBT4CBT
- Standard Treatment as Usual (TAU) (Active Comparator): Treatment that would normally be received at the clinic typically consisting of individual or group counseling sessions focusing on substance abuse.
  Interventions: Behavioral: Standard Treatment As Usual (TAU)

INTERVENTIONS:
Behavioral: Standard Treatment As Usual (TAU) — Treatment normally offered at this clinic which could include individual or group drug counseling sessions one time per week last one hour each time.
  Arms: Standard Treatment as Usual (TAU)
Behavioral: Individual clinician-provided CBT — Individual drug counseling sessions with trained clinicians using CBT one time per week last one hour per session.
  Arms: Individual clinician-provided CBT
Behavioral: CBT4CBT — Subjects work with a computerized program that teaches skills for stopping drug use and increasing coping skills. Computerized sessions are one time per week and last about one hour per session.
  Arms: CBT4CBT

SUMMARY:
The investigators are conducting a randomized clinical trial of our new web-based version of the CBT4CBT program to evaluate its effectiveness relative to standard outpatient counseling at SATU. The computer-based training program (CBT4CBT) focuses on teaching basic coping skills, presenting examples of effective use of coping skills in a number of realistic situations in video form, and providing opportunities for patients to practice and review new skills while receiving substance abuse treatment.

DETAILED DESCRIPTION:
One hundred eighty drug-using individuals seeking treatment at the Substance Abuse Treatment Unit (SATU) of the Connecticut Mental Health Center will be randomized to (1) standard outpatient counseling at SATU (typically consisting of weekly group counseling), (2) individual clinician delivered CBT, or (3) web-based CBT4CBT. Treatments will be delivered over a 12-week period with a six-month follow-up after termination of the study treatments. The primary outcome measures will be reduction in substance use (frequency of drug use by time, confirmed by urine toxicology screens). Secondary outcomes will include treatment utilization and cost, several measures intended to detect whether web-based CBT4CBT retains key characteristics of traditional clinician-administered CBT (e.g., acquisition of coping skills, use of change strategies), participant characteristics which will be evaluated as potential moderators of outcome, as well as participant satisfaction and treatment credibility.

ELIGIBILITY:
Inclusion Criteria:

* Are 18 years of age or older.
* Are applying for outpatient, non-agonist substance abuse treatment at SATU.
* Meet current DSM-IV criteria for cocaine, marijuana,opioid,or amphetamine dependence.
* Are sufficiently stable for 12 weeks of outpatient treatment.
* Can commit to 12 weeks of treatment and are willing to be randomized to treatment
* Are willing to provide locator information for follow-up.
* Are fluent in English and have a 6th grader or higher reading level

Exclusion Criteria:

* Have an untreated bipolar or schizophrenic disorder.
* Who have a current legal case pending such that incarceration during 12-week protocol is likely.
* Are physically dependent on alcohol, opioids or benzodiazepines

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Actual)
Dates: Start 2012-01; Primary Completion 2018-01 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Reduction in drug abuse | 12 weeks

SECONDARY OUTCOMES:
Subjects ability to demonstrate coping skills through a computerized role-playing evaluation | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Carroll, PhD, Principal Investigator — Yale University
Locations (1):
- Substance Abuse Treatment Unit (SATU), New Haven, Connecticut, United States

REFERENCES:
- [Derived] Kiluk BD, Nich C, Buck MB, Devore KA, Frankforter TL, LaPaglia DM, Muvvala SB, Carroll KM. Randomized Clinical Trial of Computerized and Clinician-Delivered CBT in Comparison With Standard Outpatient Treatment for Substance Use Disorders: Primary Within-Treatment and Follow-Up Outcomes. Am J Psychiatry. 2018 Sep 1;175(9):853-863. doi: 10.1176/appi.ajp.2018.17090978. Epub 2018 May 24. PMID 29792052